CLINICAL TRIAL: NCT05615961
Title: Effect of Probiotics on Endurance Athletes' Microbiome at Rest and Post-race
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Liverpool John Moores University (Other)
Collaborators: Georgia Southern University (Other); University of Illinois at Chicago (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 021/SPS/051
Record Dates: First submitted 2022-11-02; First posted 2022-11-14 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Gut Microbiome; Gut Microbiota; Aerobic Exercise; Gastrointestinal Tract Irritation; Athletes; Probiotics
Keywords: Probiotics; Endurance Exercise; Triathlon; GI Disturbance; Gut Microbiome
MeSH Terms: interventions — Probiotics

STUDY DESIGN:
Intervention Model Description: Participants are assigned into either supplement or placebo intervention groups, in a pair-matched, double-blind, placebo controlled manner.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The study has been blinded by an impartial third party from the company that has provided both the probiotic supplements and the placebo capsules.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic Supplementation Arm (Experimental): This group will receive the probiotic supplement for 4-weeks prior to their ironman race performance.
  Interventions: Dietary Supplement: Probiotics (Lab4 probiotics, Cultech, Port Talbot, Wales, UK)
- Placebo Arm (Placebo Comparator): This group will receive the placebo capsules for 4-weeks prior to their ironman race performance.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotics (Lab4 probiotics, Cultech, Port Talbot, Wales, UK) — The intervention is a unique blend of probiotic cultures from a well-established manufacturer.
  Other Names: Lab4 Probiotics, Cultech, Port Talbot, Wales, UK
  Arms: Probiotic Supplementation Arm
Dietary Supplement: Placebo — Placebo Tablets
  Arms: Placebo Arm

SUMMARY:
This study is intended to investigate the use of probiotics (LAB4 probiotics, Cultech, Port Talbot, Wales, UK) and the effect this has on gastrointestinal symptoms experienced during elite long-distance triathlon (ironman) competition, as well as the composition of the gut bacteria in the athlete.

Long-distance triathlon events frequently induce gastrointestinal discomfort due to the duration of the event (8-17 hours), the intensity of the exercise and the ingestion of large amounts of sugars throughout the event.

Data will be collected from athletes participating at the Kona ironman World-championships. Participants will supplement with either probiotic tablet, or placebo (sugar-pill) for 4-weeks prior to competition.

Athletes will be both male and female age-group athletes from any qualifying age category (age categories are as follows: 18-24; 25-29; 30-34; 35-39; 40-44; 45-49; 50-54; 55-59; 60-64; 65-69; 70-74; 75-79; 80-84).

The main investigation of the study will be the occurence/frequency/severity of gastrointestinal symptoms during training and competition between groups.

DETAILED DESCRIPTION:
The study will recruit ironman triathletes who have qualified for the Kona ironman World-championships in Hawaii. Participants will be allocated into either probiotic (Lab4 Probiotics, Cultech, Port Talbot, Wales, UK) or placebo (Maltodextrin) groups, in a double-blind fashion (Blinded by supplement supplier).

Those recruited into the study will have their training load and gut symptoms monitored for 8-weeks prior to competition via the completion of online questionnaires (previously validated).

Four-weeks prior to competition participants will provide a stool sample for microbiome analysis, they will then proceed to supplement with probiotic or placebo for 4-weeks. 24-h prior to competition they will provide a stool sample as well as providing a sample from the first bowel movement post-race, which will be used for microbiome analysis.

Data will be collected for pre-race and raceday nutrition, as well as outcome measures for raceday performance and gastroitestinal symptoms experienced, again via online questionnaire.

Stool samples will be analysed by an independent laboratory that specialises in microbiome analysis.

Primary outcome measures will be the composition of the gut bacteria and the metabolites (substances produced) of the gut bacteria at baseline, pre-race and post-race. As well as the occurrence (frequency, duration, severity) of gastrointestinal symptoms during training and competition.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-85
* Qualification for the Kona Ironman World-championships in Hawaii

Exclusion Criteria:

* Have a current musculoskeletal injury.

  * Currently unwell with cold or flu
  * Have been told they have liver disease
  * Have gastric Ulcer or other gastric/stomach problems
  * Have a condition/disease of the Gut/bowel.
  * Have diagnosed uncontrolled asthma
  * Have kidney problems
  * Have a chronic connective tissue disorder
  * Have suffered cerebrovascular disease such as a stroke
  * Are taking balcofen, methotrexate, tacrolimus and voriconazole, beta-blockers or diuretics drugs

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2022-10-10 (Actual); Study Completion 2022-10-10 (Actual)

PRIMARY OUTCOMES:
Composition of the gut microbiome | 4-weeks
  This will assess the bacterial content in the gut of the participants, performed using shotgun metagenomic sequencing
Gastrointestinal symptoms during training and competition | 8-weeks
  This will be the subjective assessment of any gastrointestinal symptoms experienced during training and competition, from a previously validated questionnaire

SECONDARY OUTCOMES:
Training volume and intensity | 8-weeks
  This will be a quantification of the amount of training completed in the 8 weeks leading up to the race, via questionnaire.
Perceived stress | 8-weeks
  This will be the subjective assessment of how stressed participants are in the 8 weeks leading up to competition, via questionnaire.
Quality of sleep | 8-weeks
  This will be a subjective assessment of how well-rested the participants are in the 8 weeks leading up to competition, via questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- Liverpool John Moores University, Liverpool, Merseyside, United Kingdom

IPD SHARING:
Plan to Share IPD: No